CLINICAL TRIAL: NCT06917040
Title: Enhancing Protection Against Vector-borne Diseases in Forcibly Displaced Communities: Evaluating the Efficacy of Spatial Repellents for Cutaneous Leishmaniasis Control in North-East Syria
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: The Mentor Initiative (Other)
Collaborators: University of Nevada, Las Vegas (Other); Hacettepe University (Other)
Responsible Party: Principal Investigator, Richard Allan, Principal Investigator, The Mentor Initiative
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CGCSR-Syria
Record Dates: First submitted 2025-04-01; First posted 2025-04-08 (Actual); Last update posted 2025-04-08 (Actual); Status verified 2025-04

CONDITIONS: Leishmaniasis, Cutaneous; Vector Borne Diseases
Keywords: Conflict; Internally displaced people; temporary shelter; spatial repellants
MeSH Terms: conditions — Leishmaniasis, Cutaneous; Vector Borne Diseases

STUDY DESIGN:
Masking Description: Neither the deliverers of the intervention nor the outcome assessors are blinded to the group allocations
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention (Experimental): 2 clusters received: 1.The study intervention was Mosquito ShieldTM. The active ingredient releases on a controlled basis over a 1-month period (1 emanator in rooms up to 18 m 2 / 2 emanator per 9 m). The households in the intervention arm were provided with Mosquito ShieldTM for 9 months (April-December 2021). This was distributed directly to households every month with pictogram instructions in the local language describing the correct intervention usage: how to open Mosquito ShieldTM, the number to be installed per room, how to attach and position Mosquito ShieldTM and the duration of Mosquito ShieldTM usage (30 days) prior to replacement. 2. IECs (brochures and posters) with information on cutaneous leishmaniasis transmission, prevention, clinical symptoms, correct treatment seeking practices and treatment locations. 3. Free of charge access to diagnostic and treatment services
  Interventions: Device: Spatial repellant emanator
- Control (No Intervention): 4 clusters received: 1. IECs (brochures and posters) with information on cutaneous leishmaniasis transmission, prevention, clinical symptoms, correct treatment seeking practices and treatment locations. 2. Free of charge access to diagnostic and treatment services

INTERVENTIONS:
Device: Spatial repellant emanator — Spatial emanator with an active ingredient Transfluthrin (C15H12Cl2F4O2, 110mg, EPA registered number 432-1588).
  Arms: Intervention

SUMMARY:
The aim of this study is to determine the efficacy of Mosquito Shield (spatial repellent) in reducing cutaneous leishmaniasis case incidence among internally displaced persons and sandfly density in temporary shelters and camp settings in Ar-Raqqa governorate, North-East Syria.

ELIGIBILITY:
Inclusion Criteria:

Known history of cutaneous leishmaniasis in camp Sleeping under same shelter type (all UNHCR tents / plastic sheets) Camp easily accessible by road Camps a minimum of 5km apart Adequate security levels

Exclusion Criteria:

Camps closer than 5km from a camp included in the study Camps with no previously recorded cases of cutaneous leishmaniasis Displaced communities living outside of defined camp settings

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 18404 (Actual)
Dates: Start 2021-02-01 (Actual); Primary Completion 2022-04-01 (Actual); Study Completion 2022-04-01 (Actual)

PRIMARY OUTCOMES:
Epidemiological outcome: cutaneous leishmaniasis incidence | 11 or 9 months
  Cutaneous leishmaniasis incidence per 1,000 will be estimated as the total number of cutaneous leishmaniasis episodes per 1,000 persons over the course of the trial. Two different incubation times or diagnostic cut-offs will be used: at 2 months post-intervention (from August 2021 to April 2022) and at 4 months post-intervention (from August 2021 to April 2022).
Entomological outcome: phlebotomine sandfly density | 9 months
  Phlebotomine sandfly density will be estimated monthly using Centers for Disease Control and Prevention light traps inside shelters.

SECONDARY OUTCOMES:
Intervention feasibility, acceptability and uptake | 11 months
  To measure community and household intervention acceptability and uptake, a questionnaire will be conducted post-intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Richard J Allan, PhD, Principal Investigator — The Mentor Initiative
Locations (1):
- The MENTOR Initiative, North East Syria, Ar-Raqqa, Syria

REFERENCES:
- [Derived] Allan R, Scherrer R, Kasap OE, Paris L, Scott T, Sauskojus H, Wetherill O, Estecha-Querol S, Alkhalaf Z, Karakus M, Yilmaz A, Alten B, Messenger LA. Enhancing protection against vector-borne diseases in forcibly displaced communities: evaluating the efficacy of spatial repellents for cutaneous leishmaniasis control in North-East Syria. BMC Med. 2025 Jul 3;23(1):401. doi: 10.1186/s12916-025-04244-2. PMID 40611204